CLINICAL TRIAL: NCT06087042
Title: Association of Serum and Salivary Dipeptidyl Peptidase-4 (DPP-4) With Oral Cancerous and Precancerous Lesions; an Observational Diagnostic Accuracy Study
Brief Title: Dipeptidyl Peptidase-4 Link With Oral Cancer and Premalignant Lesions
Status: Completed | Type: Observational
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Nayroz Tarrad, associate professor, Fayoum University
Other Study IDs: : IRB00012891#77
Record Dates: First submitted 2023-10-11; First posted 2023-10-17 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Oral Premalignant Lesions as Leukoplakia and Lichen Planus; Oral Cancer
Keywords: oral cancer; saliva; serum; dipeptidyl peptidase; potentially malignant lesions.
MeSH Terms: conditions — Lichen Planus; Mouth Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group I: patients suffering from oral squamous cell carcinoma
  Interventions: Diagnostic Test: serum and unstimulated salivary samples
- Group II: patients diagnosed with potentially malignant lesions such as leukoplakia, and dysplastic erosive or atrophic oral lichen planus
  Interventions: Diagnostic Test: serum and unstimulated salivary samples
- Group III: individuals with no oral mucosal lesions
  Interventions: Diagnostic Test: serum and unstimulated salivary samples

INTERVENTIONS:
Diagnostic Test: serum and unstimulated salivary samples — Participants were told to cease smoking, eating, or drinking before the collection of samples by about half an hour. Obtaining the sample was done by demanding the individual to swallow then incline his head forward to expectorate saliva in a sterile tube for about 3 min. Afterwards the samples were coded by serial numbers then stored at -20°C until being assessed.
  Under aseptic circumstances and using plain tubes, 5ml peripheral venous blood samples were collected from all participants by standard venipuncture. Samples were transported to biochemistry laboratory and centrifuged followed by filtration of the clarifying supernatant and then stored at -20ºC

SUMMARY:
Aim: The current study targets linking serum and salivary dipeptidyl peptidase-4 with oral squamous cell carcinoma and comparing it with potentially malignant lesions and control to validate dipeptidyl peptidase-4 as a diagnostic marker for early detection of oral cancer and to reveal its possible role in carcinogenesis.

Methodology: A total of 45 patients were recruited and subdivided into 2 groups: Group I: 15 patients having oral squamous cell carcinoma. Group II: 15 patients with potentially malignant lesions (leukoplakia and oral lichen planus) compared to 15 systemically healthy participants having no oral mucosal lesions acting as a control group (Group III). Serum and whole unstimulated salivary samples were collected from all participants to evaluate dipeptidyl peptidase level in different groups using enzyme linked immune-sorbent assay (ELISA) kit. ROC analysis was done to reveal area under the curve, sensitivity, specificity and diagnostic accuracy of DPP-4 among different groups.

ELIGIBILITY:
Inclusion Criteria:

* systemically healthy
* No current medication,
* both genders with age ranging from 30 to 65 years old.
* having oral leukoplakia, oral lichen planus or oral squamous cell carcinoma

Exclusion Criteria:

* systemic disease
* pregnancy
* lactation
* being diagnosed with any other oral mucosal lesion

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: adult individuals entering in the out patient clinics of oral medicine and diagnosis department
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2023-08-15 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
DPP-4 level detection | level of DPP-4 is measured after the completion of all sample collection carried at the day of enrollment of subjects in the investigation after diagnosis confirmation
  level of DPP-4 is measured in all collected serum and salivary samples

CONTACTS AND LOCATIONS:
Overall Officials: Nayroz Tarrad, associate professor, Principal Investigator — faculty of dentistry, Fayoum university
Locations (1):
- faculty of dentistry, Fayoum university, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abdel Fattah Tarrad N, Gamil Shaker O, Abdelkawy M, Hassan S. Association of serum and salivary dipeptidyl peptidase-4 (DPP-4) with oral cancerous and precancerous lesions; an observational diagnostic accuracy study. BMC Oral Health. 2024 Oct 10;24(1):1206. doi: 10.1186/s12903-024-04939-7. PMID 39390508